CLINICAL TRIAL: NCT04560127
Title: A Single-arm, Non-randomized, Single-center Study to Evaluate Camrelizumab in Combination With Apatinib in Patients With Radioactive Iodine-refractory Differentiated Thyroid Cancer
Brief Title: Camrelizumab in Combination With Apatinib in Patients With Radioactive Iodine-refractory Differentiated Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yansong Lin, Vice-director, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-TC-II-003/Ahead-T204
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Radioactive Iodine-refractory Differentiated Thyroid Cancer
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Camrelizumab combination with Apatinib (Experimental): Apatinib (250mg p.o. q.d.) combined with Camrelizumab (200mg, iv, q2w)
  Interventions: Drug: Camrelizumab combination with Apatinib

INTERVENTIONS:
Drug: Camrelizumab combination with Apatinib — Apatinib (250mg p.o. q.d.) combined with Camrelizumab (200mg, iv, q2w)

SUMMARY:
This is a single arm, open-label, non-randomized and single-center phase II clinical study, to evaluate the safety, tolerance, and efficacy of Camrelizumab in combination with Apatinib in patients with Radioactive Iodine-refractory Differentiated Thyroid Cancer (RAIR-DTC).

DETAILED DESCRIPTION:
It is estimated that 10 patients who met the study criteria will be enrolled in 1 years and treated with Camrelizumab plus Apatinib in PUMCH. The investigators will follow up and collect subjects' data to evaluate the efficacy and safety of treatment, including objective response rate (ORR) and Progression-free Survival (PFS) and Overall Survival (OS), until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

1. Aged after 18 years (18 is included). 2. Locally advanced or metastatic differentiated thyroid cancer (papillary, follicular, Hurthle cells, poorly differentiated carcinoma). At least one measurable lesion (helical CT scan long diameter ≥10mm, meet the requirements of the standard Response Evaluation Criteria In Solid Tumors（RESCIST） version 1.1).

3. ECOG-PS score 0-2 4. Life Expectancy of at least 12 weeks 5. Subjects must be 131I-refractory / resistant as defined by at least one of the following.

1. Lesions that do not demonstrate iodine uptake on any radioiodine scan.
2. Subjects received a single radioactive iodine therapy within 12 months (≥ 3.7 Giga Bequerel（GBq）[≥ 100 millicurie（mCi）]) and target lesion disease progression.
3. Every two radioactive iodine treatment interval <12 months, doses ≥ 3.7 GBq [≥100mCi], disease progress more than 12 months after at least once iodine therapy.
4. Received a total dose of radioactive iodine therapy ≥ 22.2 GBq (≥ 600 mCi). 6. Have the required screening laboratory values.

Exclusion Criteria:

1. Other thyroid cancer histological subtypes (such as medullary carcinoma, lymphoma or sarcoma).
2. Any active autoimmune disease or history of autoimmune disease and expected recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis); subjects with skin diseases that does no need systemic treatment, for example, leukoderma, psoriasis, alopecia, those with controlled type I diabetes by insulin or those with asthma that has been completely resolved in childhood and with no need of any intervention can be enrolled; while subjects with asthma who need bronchodilator for medical intervention cannot be enrolled.
3. Use of strong CYP3A4/CYP2C19 inducers, including rifampicin (and its analogues) and St. John's Wort, or strong CYP3A4/CYP2C19 inhibitors within two weeks prior to signing informed consent form.
4. Previous treatment with other immune checkpoint inhibitors (include PD-1 antibody or other immunotherapy against PD-1/PD-L1).
5. Known history of serious allergy to any monoclonal antibody or Apatinib.
6. Inability or unwilling to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption.
7. Previous or current presence of metastasis to central nervous system.
8. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia or complications of severe pneumonia; oral or intravenous therapeutic antibiotics within two weeks prior to the start of study treatment (for example, subjects who are given with preventive antibiotics for prevention of urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible for participation in the study).
9. Pregnant or lactating women.
10. Other factors that may affect the study results or lead to forced termination of the study early as judged by investigators, such as alcoholism, drug abuse, other serious diseases (including mental disorders) requiring concomitant therapy, with serious laboratory examination abnormality, with family or social factors, that may affect subject's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time Frame: two years
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.

SECONDARY OUTCOMES:
Overall Survival (OS) | two years
  Duration from the date of initial treatment to the date of death due to any cause.
Progression-free Survival (PFS) | two year
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1) or death of any cause.
Disease Control Rate (DCR) | two year
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Duration of Response (DoR) | two year
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Time to Progression (TTP) | two year
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1)
Adverse events (AE) | two years
  Any adverse events related with treatment drugs and details include adverse events type, frequency and severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Sun D, Zhang Y, Mu Z, Shi C, Sun Y, Cheng X, Meng C, Wei X, Liang J, Lin Y. Camrelizumab and apatinib in Chinese patients with locally advanced or metastatic radioiodine-refractory differentiated thyroid cancer: an exploratory open-label, single-arm trial. BMC Med. 2025 Dec 18. doi: 10.1186/s12916-025-04550-9. Online ahead of print. PMID 41408254